CLINICAL TRIAL: NCT01856335
Title: Increasing Self-Efficacy and Outcome Expectations For Exercise in Adults With Epilepsy: An Educational Motivation Intervention - E-MOVE
Brief Title: Exercise Education for Adults With Seizure Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 130127; 13-N-0127
Record Dates: First submitted 2013-05-10; First posted 2013-05-17 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12-07

CONDITIONS: Seizures; Epilepsy
Keywords: Seizures; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Patient Education as Topic

INTERVENTIONS:
Other: Patient Education
Other: exercise: increase physical activity/goal setting

SUMMARY:
Study Population

-People with seizures benefit from regular exercise. Exercise may help decrease the number of seizures they have. It also improves overall health and quality of life. However, people with seizure disorders often have been prevented from doing sports or other regular physical activity. They may also feel that exercise or injury can increase their risk of seizures. Researchers want to try an exercise program for people who have seizures to see if they can increase motivation to exercise which will improve overall health and may decrease the frequency of seizures.

Objectives:

- To see how exercise education improves motivation to exercise in people who have a history of seizures.

Eligibility:

- Individuals at least 18 years of age who have a history of seizures.

Design:

* This study involves three outpatient visits and weekly telephone calls for about 12 weeks. There will be followup calls at about 6 and 12 months after the outpatient visits.
* Participants will be screened with a physical exam and medical history. They will answer questions about their current level of physical activity, mood, quality of life, and ideas about exercise.
* At the first visit, participants will learn how to keep a physical activity log and seizure calendar. They will also use an activity monitor and take their pulse regularly. They will complete questionnaires about their mood and thoughts about exercise and seizures.
* At the second visit, participants will set personal activity goals and learn about physical activity and seizures. They will review the physical activity log, seizure log, and activity monitor and pulse readings for the previous 4 weeks.
* After the second visit, participants will receive weekly telephone calls. Each call will last about 5 minutes. These calls will ask about physical activities for the week and participants' progress toward meeting their goals. These calls will also review the seizure log.
* At the third visit (12 weeks), the same tests from the first visit will be repeated.
* The followup phone calls will continue to monitor participants' activity levels.

DETAILED DESCRIPTION:
Objective:

To see what keeps people with seizures from exercising and see how they can increase their belief that they can exercise and that exercise will help them.

Study Population:

50 adults with seizures

Design:

In this protocol, we will pilot the use of an educational intervention to provide people with seizure disorders an opportunity to learn about the benefits of exercise and learn specifically what types of exercise to incorporate into their daily lives.

Outcome Measures:

To assess the effectiveness of the educational intervention, we will use pre and post intervention measures including seizure specific measures of self-efficacy (belief that they can exercise) and outcome expectations (belief that exercise will help them) for exercise. To assess changes in physical activity, seizure frequency, and mood, we will monitor physical activity and seizure calendars, activity monitor recordings, and mood rating scales.

ELIGIBILITY:
* INCLUSION CRITERIA:

Able to use seizure calendars to record seizures throughout the study

English speaking

Able to provide informed consent

Diagnosed with epilepsy by standard clinical criteria.

Age 18 years and older

Enrolled in evaluation and treatment of epilepsy protocol 01-N-0139

EXCLUSION CRITERIA:

Do not have health care provider clearance to participate in a physical activity program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05-10; Primary Completion 2017-01-25 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Change in Self-efficacy for exercise score following the E-MOVE intervention. | 0 and 12 weeks post intervention
Change in Outocme Expectations for exercise score following the E-MOVE intervention. | 0 and 12 weeks post intervention

SECONDARY OUTCOMES:
The effect of the E-MOVE intervention on seizure frequency based on seizure calendar self-report, quality of life scores, symptoms of depression and BMI measures. | 0 and 12 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Irene H Dustin, C.R.N.P., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arida RM, Cavalheiro EA, da Silva AC, Scorza FA. Physical activity and epilepsy: proven and predicted benefits. Sports Med. 2008;38(7):607-15. doi: 10.2165/00007256-200838070-00006. PMID 18557661
- [Background] Arida RM, Scorza CA, Schmidt B, de Albuquerque M, Cavalheiro EA, Scorza FA. Physical activity in sudden unexpected death in epilepsy: much more than a simple sport. Neurosci Bull. 2008 Dec;24(6):374-80. doi: 10.1007/s12264-008-0805-z. PMID 19037323
- [Background] Arida RM, Scorza FA, Cavalheiro EA. Favorable effects of physical activity for recovery in temporal lobe epilepsy. Epilepsia. 2010 Jul;51 Suppl 3:76-9. doi: 10.1111/j.1528-1167.2010.02615.x. PMID 20618406